CLINICAL TRIAL: NCT01816568
Title: The Comparison of Single Incision Laparoscopic Appendectomy and Three Port Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, manuk norayk manukyan, Assoc.Prof., Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mütf4
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Acute Appendicitis
Keywords: appendicitis, laparoscopy, single incision
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): SILS appendectomy
  Interventions: Procedure: SILS appendectomy
- Group 2 (Active Comparator): Three port laparoscopic appendectomy
  Interventions: Procedure: Three port laparoscopic appendectomy

INTERVENTIONS:
Procedure: SILS appendectomy — Single incision laparoscopic appendectomy will be performed
  Arms: Group 1
Procedure: Three port laparoscopic appendectomy — Three port laparoscopic appendectomy will be performed
  Arms: Group 2

SUMMARY:
Laparoscopic techniques have allowed surgeons to perform complicated intrabdominal surgery with minimal trauma. In numerous studies, when conventional laparoscopic appendectomy using 3 ports is compared with open appendectomy, it has advantages of reduced pain, reduced hospital stay, and enhanced cosmetic effects. Single incision laparoscopic surgery (SILS) was developed with the aim of reducing the invasiveness of conventional laparoscopy. In this study the investigators aimed to compare results of SILS appendectomy and three port conventional laparoscopic appendectomy prospectively.

DETAILED DESCRIPTION:
Total of 50 patients who undergoing laparoscopic appendectomy for acute appendicitis will randomly assign to undergo SILS appendectomy group (n = 25) or Three port laparoscopic appendectomy group (n= 25) according to a computer-generated table of random numbers. Demographics (ie, age, gender, body mass index (BMI), American Society of Anesthesiology (ASA) score, need for conversion to a standard or three port laparoscopic appendectomy, need for conversion to an open appendectomy will be recorded. Outcome measures include operative morbidity, operative time, pain score, hospital stay. Morbidity will be evaluated by rates of colonic leak, wound infection, intrabdominal abscess hospital readmission, and hernia.

ELIGIBILITY:
Inclusion Criteria:

* Required laparoscopic cholecystectomy for gallbladder disease.

Exclusion Criteria:

* American Society of Anesthesiologists score (ASA) more than III,
* Patients had prior abdominal surgery,
* Pregnancy,
* Ongoing peritoneal dialysis,
* Lack of written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pain score | Postoperative first 24 hours
  Postoperative pain will be assessed according Visual analog scale from 0 (no pain) to 10 (worst pain imaginable. Postoperative six hour VAS (POSH-VAS) and postoperative first day VAS (POFD-VAS) will be recorded and compared.

SECONDARY OUTCOMES:
Intraoperative complications | Average of 50 minutes
  Per operative complications will be recorded.
  * Bleeding
  * Iatrogenic injury
  * Bowel perforation
  * Complications associated with increased intra-abdominal pressure
Operating time | Average of 50 minutes
  The operating time will be defined as the time from the first incision to the last suture's placement.
Postoperative complications | 24th hour, 2nd day, 3rd day, 7th day, 1st month, 3rd month, 6th month, 1st year
  Postoperative complications will be recorded postoperative follow up.
  * Bleeding
  * Fecal leakage
  * Intrabdominal injury
  * Wound infection
  * Port site hernia

OTHER OUTCOMES:
Length of hospital stay | Average of 2 days
  Length of hospital stay will be recorded postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Deveci, Assoc.Prof., Principal Investigator — Maltepe University School of Medicine, General Surgery Department; Fatih Altintoprak, Assoc.Prof., Principal Investigator — Sakarya University School of Medicine, General Surgery Department; Manuk Norayk Manukyan, Assoc.Prof., Study Director — Maltepe University School of Medicine, General Surgery Department; Sertan Kapakli, Assoc.Prof., Principal Investigator — Maltepe University School of Medicine, General Surgery Department; Abut Kebudi, Prof., Study Chair — Maltepe University School of Medicine, General Surgery Department